CLINICAL TRIAL: NCT07193446
Title: Optimising the Delivery of Diabetes Distress Informed Care for Its Prevention, Detection, and Management in Adults With Type 1 Diabetes: a Feasibility Study (D-stress Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 349849; PGfAR NIHR205441 (Other Grant/Funding Number: National Institute of Health Research (NIHR))
Record Dates: First submitted 2025-08-13; First posted 2025-09-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): This arm of the study involves health care professionals e-learning training in and delivery of EUC for the detection and management of diabetes distress.
  Interventions: Behavioral: D-stress study: The detection, prevention and management of diabetes distress for adults living with type 1 diabetes.
- REDUCE Programme Intervention (Experimental): REDUCE intervention is an online group 6 session programme for the management of elevated diabetes distress.
  Interventions: Behavioral: D-stress study: The detection, prevention and management of diabetes distress for adults living with type 1 diabetes.

INTERVENTIONS:
Behavioral: D-stress study: The detection, prevention and management of diabetes distress for adults living with type 1 diabetes. — Enhanced Usual Care intervention aims to train health care professionals to detect and prevent, and manage diabetes distress in routine diabetes care, in the UK NHS. The REDUCE programme aims to prevent and manage elevated diabetes distress.

SUMMARY:
Up to one in two adults with type 1 diabetes find living with and managing diabetes to be emotionally challenging. This 'emotional side' of diabetes - feeling worried, frustrated, overwhelmed, sad, burnt-out - is called diabetes distress. It affects people's quality of life and can hinder them from managing their diabetes as well as they can.

In the UK, the NHS needs to better understand how to best support people feeling emotionally burdened by diabetes. So, we have worked with diabetes distress specialists around the world to develop an NHS pathway to care for diabetes distress. This pathway to care involves training diabetes teams to recognise, assess and talk about diabetes distress at routine appointments. If people have a high diabetes distress level, they may be able to take part in an online group program to help them manage their type 1 diabetes and emotions. The feasibility study will test this pathway to care with people with type 1 diabetes in the NHS setting.

ELIGIBILITY:
Inclusion Criteria:

Adults with type 1 diabetes

* People aged 18 years old and older
* With a T1DM diagnosis of more than one year
* Who used a Continuous Glucose Monitoring device 3 months prior to trial entry

Health care professionals

* Members of the multidisciplinary diabetes team
* Who would like and be able to undertake training in Enhanced Usual Care (EUC)

Family or friend

* People aged 18 years or older
* Is involved with the care of the participant
* The participant has consented to the family member or friend to be involved in the study

REDUCE Facilitators

• Eligibility as per the role specification in Section 6.2.2 of study Protocol

Exclusion Criteria:

Adults with type 1 diabetes

* Exclusion criteria will include those adults diagnosed less than one year ago. This is because the first 12 months following a diagnosis of T1DM is a period of unique stress due to the diagnosis, the acute onset, and requirement to learn complex new skills. Additionally, due to the honeymoon period, which can typically last up to a year, there is variety in the physiological trajectory which might have an impact that would be difficult to measure and account for in this study(Sokołowska, Chobot et al. 2016).
* Women who are pregnant. This is because the additional burdens and anxieties this population is confronted with may risk confounding the trial findings
* Exclusion of adults with current mental health diagnoses with current symptoms (e.g. psychosis or substance abuse or severe depression), will be evaluated and determined on a case-by-case basis by clinical care teams.

Health care professionals • People who are unwilling or unable to take on additional workload associated with D-stress e-learning and delivery of Enhanced Usual Care.

Family or friend

• Participant with type 1 diabetes has not given consent for a family member or friend to participate in the study

REDUCE Facilitators

* • Professional accreditation with one of the following professional bodies: Nursing & Midwifery Council, Health & Care Professionals Council, British Association for Counselling & Psychotherapy, and UK Council for Psychotherapy.
* Professional or personal understanding of Type 1 diabetes
* Professional or personal understanding of NHS diabetes care and guidelines
* Professional or personal understanding of diabetes distress
* Professional understanding of mental and emotional health
* Professional experience of in-person and/or online group facilitation especially in managing diverse needs within a group and the expression of strong emotions
* Willingness to be a research participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility, service use, acceptability, attrition rate and data quality | The study investigators will be collecting data to assess the primary outcome measure at Month 3 and Month 6 of the study.
  The main primary outcome measure is to assess the feasibility of the study in relation to progressing to the proposed main trial. As part of the primary outcome the study investigators will be assessing the following:
  1. Extent to which of participants find the interventions feasible, and acceptable
  2. Proportion of people recruited from those eligible/approached
  3. The number of participants who dropped out
  4. The quality of the data To conduct these assessments measurements tools used will include: the Acceptability, feasibility and appropriateness of implementation (AIM) (Sturt, Griffiths et al. 2023; Weiner, Lewis 2017), and EQ-5D-5L Quality of Life questionnaire (Feng, Kohlmann et al. 2021). The AIM and EQ-5D-5L measurement tools uses a Likert scale as a unit of measure.
Diversity of recruited participants against nine protected characteristics | This primary outcome data will be collected at month 3 baseline data collection and month 6 follow-up data collection.
  The study investigators will be assessing the diversity of recruited participants against against nine protected characteristics with the D-stress study specific measurement tool called, the Health and social equalities.
To assess the quality of data collected | The study investigators will be collecting data to assess the primary outcome measure at monthly throughout the duration of the 6 month study.
  As part of the primary outcome the study investigators will be assessing the quality of data collected via monthly questionnaires using the Acceptability, feasibility and appropriateness of implementation (AIM) (Sturt, Griffiths et al. 2023; Weiner, Lewis 2017), measurement tool realist evaluation process interviews and non-participant observation with study investigators following RAMESES quality and publication standards guidelines (Wong G, Greenhalgh T, Westhorp G, et al. 2013).

SECONDARY OUTCOMES:
Assessment of initial Realist Process Evaluation programme theories | Conducted over the course of the feasibility study from Day 1 through to the completion of the study, an average of 6 months.
  Assessing whether the initial programme theories underpinning Enhanced Usual Care (control) and REDUCE programme (experimental) explain the outcomes and participant experiences of these interventions. Non-participant observations of control and experimental intervention will be conducted. Realist Process Evaluation interviews with study participants will also be conducted over the course of the study: from day 1 (month 1) through to month 6.
Proportion of TIR for interstitial blood glucose (proposed main trial co-primary outcome) | CGM data will be collected monthly from Month 1 through to study completion, an average of 6 months.
  The proportion of time interstitial blood glucose is in the range of 4-10 mmol/l (Battelino, Alexander et al. 2022). This will be collected via the participant's continuous glucose monitoring (CGM) device every 30 days (each month) from the start of the study (month 1) through to study completion, an average of 6 months.
  In addition to proportion of time interstitial blood glucose is in the range , below range, above range, and glucose variability, measured as coefficient of variation will be measured. Percentage of CGM sensor usage will also be measured. This will allow study investigators to determine the completeness of interstitial blood glucose sensor data and proportion of time in the preceding month the participant's blood glucose was in range.
Diabetes distress score (proposed main trial co-primary outcome) | The T1-DDAS measurement scale will be used every 30 days from Month 1 through to study completion, estimated to be 6 months.
  The Type 1 Diabetes Distress Assessment Scale T1-DDAS 8-item CORE scale will be the key scale used to collect diabetes distress levels. Items are scored between 1 and 5, with one being Not a problem to five being A very serious problem. A core score of under 3 on each item is sub-threshold and ≥3 is elevated. The tool was 'developed and validated and standardized' for adults with Type 1 diabetes by the Behavioural Diabetes Institute to further specify the source of DD as well as the amount of DD (Institute, 2023; Fisher, Polonsky et al. 2024).

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal United Hospitals Bath, Bath
  - University Hospitals Leicester NHS Trust, Leicester
  - Guy's and St Thomas' Hospitals NHS Trust, London